CLINICAL TRIAL: NCT00969995
Title: Identification of Inflammatory Markers in Migraine Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Amnon Mosek, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-AM-197-CTIL
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Inflammation; Migraine; Headache
Keywords: inflammation; migraine; headache
MeSH Terms: conditions — Inflammation; Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- migraine1: 50 subjects with migraine without aura
- migraine 2: 50 subjects with migraine with aura
- tension: 50 subjects with tension headache
- cluster: 50 subjects with cluster headache
- Healthy: 50 healthy subjects

SUMMARY:
Migraine is prevalent in 10-12% of the population. It involves the development of a cranial perivascular neurogenic inflammation. Recent information suggests that migraine might be a risk factor to stroke. The possible mechanisms that might relate migraine and stroke are: 1. Migraineous infarction 2. A primary endothelial disorder. 3. Genetic relation 4. An ongoing inflammatory process. C reactive protein (CRP) is a sensitive marker for an inflammatory process.The data on the relation of migraine to inflammation is limited. The aim of the current study is to assess inflammatory factors as possible markers for migraine.

DETAILED DESCRIPTION:
Migraine is prevalent in 10-12% of the population, with female preponderance (1). Migraine may cause a significant distress and reduction of the quality of life of the patients, of whom in almost a third of them the migraine attack reduces the ability to function. The main form of migraine is migraine without aura while 20-30% of the patients have migraine with aura (2) which is a focal neurological phenomenon that occurs 20-30 minutes prior to the migraine pain. The development of a cranial perivascular neurogenic inflammation hallmarks the migraine attack which involves the secretion of vasodilatatory and inflammatory peptides from the perivascular intracranial trigeminal terminals (3).

Recent information suggests that migraine might be a risk factor to stroke. Migraineurs were found to carry a higher risk to develop stroke when compared to subject without migraine, and this risk was higher among patients with migraine with aura (4-6) and in particular in women 45 years of age or younger (7-8). Brain MRI studies showed that migraineurs have more sub-clinical infarcts and abnormal white matter signals, in particular among young women with migraine with aura compared to normal controls (9-10). Furthermore, the findings in a large prospective study suggest that the possible relation between migraine and vascular disorders is even larger, showing that patients with migraine with aura carry a higher risk to develop stroke but also myocardial infarction, compared to those who do not suffer from migraine (11). The mechanisms that relate migraine to stroke are unknown. The possible mechanisms that might relate migraine and stroke are:

1. The pathophysiological vascular changes that occur during migraine are the direct (migraineous infarction) or indirect cause of stroke (12).
2. Migraineurs have a primary endothelial disorder which could be expressed in several vascular aspects such as migraine, stroke, Renauld's phenomenon and PFO.
3. Migraine and stroke are genetically related as in familial hemiplegic migraine.
4. Migraine is accompanied by, or the cause of, an ongoing inflammatory process which is the cause of stroke (13).

C reactive protein (CRP) is a sensitive marker for an inflammatory process, rising quickly in response to an inflammation or tissue damage. CRP in not only a marker but also involved in the identification of pathogens, activation of the complementary system and phagocytic response and, therefore, has an important role in the protection from infections (14). It also has a role in the restoration of the structure and activity of damaged tissues (15). On the other hand, high levels of CRP were related to higher risk to develop a cardiovascular disease or stroke (16, 17). CRP might be a primary risk factor for these disorders (18, 19) possibly through inflammatory or hypercoagulability mechanisms (20, 21). Nevertheless, no significant correlation was found between CRP and atherosclerosis.

The data on the relation of migraine to inflammation is limited. In a retrospective study, with no control group, data on patients considered with a complicated medical problem by a neurologist were collected from the patients' files. Out of 60 patients with migraine (50% migraine with aura) 43% had high CRP levels (>3mg%; in 55% of those with migraine without aura and in 32% of those with migraine with aura) (22). A prospective study of 50 migraineurs (64% with aura) found a significantly higher CRP levels in the migraine group compared to the controls and, as the previous study, those with migraine without aura had higher levels of CRP (23). These findings possibly point on a relation between migraine and inflammation.

Aim of the study

To examine values of a 'baseline inflammatory profile' in patients with migraine with and without aura in comparison to control groups in order to identify an inflammatory marker.

A. Main study objective: to evaluate if the levels of inflammatory markers in patients with migraine is higher compared to the levels of these markers in the control groups.

B. Secondary study objective: to evaluate the levels of inflammatory markers in-between migraine and other forms of headaches.

ELIGIBILITY:
Inclusion criteria:

1. Men or women older than 18 years of age.
2. Diagnosed with migraine, tension type headache or cluster headache according to International Headache Society criteria (24).
3. Headache duration is at least 1 year prior to study entry.
4. The frequency of migraine or tension type headache is 1-6 attacks in one month. Cluster headache duration is 2-4 weeks every year.
5. No prior history of cerebral or cardiac vascular event.

Exclusion criteria:

1. Pregnant or breast feeding women.
2. Subjects with permanent treatment with steroids.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patient group will consist of 200 subjects with various headache types treated at the headache clinic at the Sourasky Medical Center, Tel-Aviv, ISRAEL, and 50 healthy controls.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate if the levels of inflammatory markers in patients with migraine is higher compared to the levels of these markers in the control groups. | 1.5 years

SECONDARY OUTCOMES:
To evaluate the levels of inflammatory markers in-between migraine and other forms of headaches. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amnon mosek, Principal Investigator — The Headache and Facial pain Clinic, the departement of Neurology, Sourasky Medical Center, Tel Aviv
Locations (1):
- The headache clinic, Sourasky Medical Center Tel Aviv, Tel Aviv, Israel